CLINICAL TRIAL: NCT00115648
Title: Extended Infant Post-exposure Prophylaxis With Antiretrovirals to Reduce Postnatal HIV Transmission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Michael Thigpen, Medical Officer, Centers for Disease Control and Prevention
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PEPI-Malawi
Record Dates: First submitted 2005-06-23; First posted 2005-06-24 (Estimated); Last update posted 2014-03-07 (Estimated); Status verified 2014-03

CONDITIONS: HIV Infections
Keywords: HIV; MTCT; Infants; africa; HIV Seronegativity
MeSH Terms: conditions — HIV Infections | interventions — Nevirapine; Zidovudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Active Comparator): Single dose NVP + ZDV daily for the first week.
  Interventions: Drug: Nevirapine; Drug: AZT; Drug: NVP and AZT
- C (Experimental): Arm A plus NVP + ZDV daily to age 14 weeks.
  Interventions: Drug: Nevirapine; Drug: AZT; Drug: NVP+AZT
- B (Experimental): Arm A plus oral NVP daily to age 14 weeks.
  Interventions: Drug: Nevirapine; Drug: NVP

INTERVENTIONS:
Drug: Nevirapine — Oral NVP daily dosage
Drug: AZT — Oral AZT daily
  Other Names: Zidovuidne (ZDV)
  Arms: A; C
Drug: NVP and AZT — Oral single dose NVP plus oral daily AZT during the first weeks
  Other Names: Nevirapine and zidovudine
  Arms: A
Drug: NVP — Oral NVP daily to age 14 weeks
  Other Names: Nevirapine
  Arms: B
Drug: NVP+AZT — Oral NVP daily plus oral AZT daly to age 14 weeks
  Other Names: Nevirapine plus zidovudine
  Arms: C

SUMMARY:
The purpose of this study is to determine if extended antiretroviral regimens given to the infant during the first 14 weeks of age would decrease breast milk transmission of HIV.

DETAILED DESCRIPTION:
This is a three-arm randomized, open label, clinical trial to evaluate the effectiveness of two extended regimens of antiretrovirals compared to infant single dose nevirapine plus AZT given twice daily for 1 week (comparison regimen). All infants receive the comparison regimen at birth and then randomized at birth to start either one of the two extended regimens after the first week. The extended regimens are nevirapine daily and nevirapine plus AZT daily - both regimens are given up to age 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Had given birth within the last 24 hours
* Ability and willingness to give informed consent for HIV testing and enrollment into the study
* Willing to receive HIV results
* HIV infected
* Planning to deliver or had given birth at the study clinics
* Willing to come back for follow-up visits for 2 years postnatally
* Resident of Blantyre city or its suburbs

Exclusion Criteria:

* HIV negative
* Women with discordant HIV results
* Women who indicate that they will not breastfeed at time of delivery
* Inability or unwillingness to follow any of the inclusion requirements
* Newborn with life-threatening condition
* Women who previously enrolled in this study and have a second pregnancy cannot reenroll

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3300 (Estimated)
Dates: Start 2004-04; Primary Completion 2007-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
A. Rate of HIV infection at 9 months and assess HIV infection rates at 6-8 & 14 weeks, and 6, 12, 18, and 24 months. B.Determine HIV survival rates at ages 6, 12, 18, and 24 months. C. Evaluate safety of oral NVP and ZDV for 14 weeks. | 9 months

SECONDARY OUTCOMES:
To determine overall infant survival rates at 6, 12, 18 and 24 months. | 6,12,18 & 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Taha E Taha, MD PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- College of Medicine, Blantyre, Malawi

REFERENCES:
- [Derived] Schwartz SR, Kumwenda N, Kumwenda J, Chen S, Mofenson LM, Taylor AW, Fowler MG, Taha TE. Maternal Highly Active Antiretroviral Therapy and Child HIV-Free Survival in Malawi, 2004-2009. Matern Child Health J. 2016 Mar;20(3):542-9. doi: 10.1007/s10995-015-1852-5. PMID 26525557
- [Derived] Redd AD, Wendel SK, Longosz AF, Fogel JM, Dadabhai S, Kumwenda N, Sun J, Walker MP, Bruno D, Martens C, Eshleman SH, Porcella SF, Quinn TC, Taha TE. Evaluation of postpartum HIV superinfection and mother-to-child transmission. AIDS. 2015 Jul 31;29(12):1567-73. doi: 10.1097/QAD.0000000000000740. PMID 26244396
- [Derived] Taha TE, Li Q, Hoover DR, Mipando L, Nkanaunena K, Thigpen MC, Taylor A, Kumwenda J, Fowler MG, Mofenson LM, Kumwenda NI. Postexposure prophylaxis of breastfeeding HIV-exposed infants with antiretroviral drugs to age 14 weeks: updated efficacy results of the PEPI-Malawi trial. J Acquir Immune Defic Syndr. 2011 Aug 1;57(4):319-25. doi: 10.1097/QAI.0b013e318217877a. PMID 21423025
- [Derived] Kumwenda NI, Hoover DR, Mofenson LM, Thigpen MC, Kafulafula G, Li Q, Mipando L, Nkanaunena K, Mebrahtu T, Bulterys M, Fowler MG, Taha TE. Extended antiretroviral prophylaxis to reduce breast-milk HIV-1 transmission. N Engl J Med. 2008 Jul 10;359(2):119-29. doi: 10.1056/NEJMoa0801941. Epub 2008 Jun 4. PMID 18525035